CLINICAL TRIAL: NCT02807571
Title: Office Based Hand Surgery Using WALANT (Wide Awake Local Anesthesia No Tourniquet): Outcomes and Cost Savings Analysis
Acronym: WALANT
Status: Withdrawn | Type: Observational
Why Stopped: Study underwent major protocol changes prior to planned enrollment
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-263
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Surgery
Keywords: Hand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Wide Awake Local Anesthesia No Tourniquet — Wide Awake Local Anesthesia No Tourniquet for office based hand surgery.

SUMMARY:
This study is aimed at determining if office based surgery is an effective way of cutting health care cost while maintaining patient safety and satisfaction.

DETAILED DESCRIPTION:
The study is a retrospective chart review with prospective patient satisfaction and functional outcome surveys.

Patients that have had office based procedures that otherwise could be performed in the outpatient surgical setting from January 1, 2015 to December 4, 2015 will be contacted for study enrollment. Patient satisfaction and functional outcome surveys will be administered to those patients that consent to the research study.

The data to be collected will include but is not limited to: age gender limb dominance, complications and co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen for office based procedures that otherwise would be performed in the outpatient surgical setting from January 1, 2015 to December 4, 2015

Exclusion Criteria:

* K-wire hardware removal
* Closed reductions
* Patients receiving antibiotics at the time of the procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients seen for office based procedures that otherwise would be performed in the outpatient surgical setting from January 1, 2015 to December 4, 2015.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Complication Rates | 2 months
  Collect the incidence of complications.

SECONDARY OUTCOMES:
Cost savings | 2 months
  Compare the costs of the WALANT procedure with similar procedures done at an ASC or as an outpatient.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jebson, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No